CLINICAL TRIAL: NCT05147870
Title: Whether Peritoneal Irrigation Intra-operatively Effects on the Outcome After Laparoscopic Surgery for Peptic Ulcer Perforation
Brief Title: Outcome After Laparoscopic Surgery for Peptic Ulcer Perforation
Status: Completed | Type: Observational
Sponsor: Chang Wei-Jung (Other)
Responsible Party: Sponsor-Investigator, Chang Wei-Jung, Sponsor-Investigator, Changhua Christian Hospital
Organization: Changhua Christian Hospital (Other)
Other Study IDs: 201021
Record Dates: First submitted 2021-11-05; First posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Intraabdominal Abscess After Procedure; Leakage; Pneumonia; Operation Wound; Infection
Keywords: Laparoscopic surgery; Perforated peptic ulcer; Peritoneal irrigation; Gauze wiping and suction; Intra-abdominal abscess
MeSH Terms: conditions — Pneumonia; Surgical Wound Infection; Peptic Ulcer Perforation; Abdominal Abscess | interventions — Peritoneal Lavage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Irrigation group
  Interventions: Procedure: Peritoneal irrigation
- Suction only group
  Interventions: Procedure: Suction only

INTERVENTIONS:
Procedure: Peritoneal irrigation — For patients allocated to the irrigation group, peritoneal lavage was performed at the surgeon's discretion based on surgical findings and preference.
  Groups: Irrigation group
Procedure: Suction only — In the suction only group, one surgical gauze each was placed in the splenophrenic space and Morison's pouch to soak up any remaining purulent fluid followed by turning the patient into the Trendelenburg position for inspection of the lower abdominal cavity. Any interloop adhesions were carefully divided and the gauze-wiping maneuver was used to soak up the residual peritoneal fluid, and all bowel loops were investigated to the root of the mesentery.
  Groups: Suction only group

SUMMARY:
Despite advances in laparoscopic surgery for perforated peptic ulcer (PPU), intra-abdominal abscess (IAA) is recognized as one of the commonly reported complications with relation to the extent of infectious abdominal contamination. Herein, the investigators report their experience of laparoscopic surgery for PPU with/without peritoneal irrigation and discuss postoperative outcome. The investigators retrospectively examined the electronic medical records of the patients who underwent laparoscopic surgery for perforated peptic ulcer at a single medical center in Taiwan between January 2013 and August 2021. Retrospectively, the investigators would include those patients with clinical diagnosis of PPU who underwent emergent laparoscopic surgery. The patients with previous abdominal surgery, pathologic confirmed malignant ulcer perforation or concomitant ulcer bleeding were excluded. The investigators focused on post-operative complications and outcome after laparoscopic surgery with or without peritoneal irrigation. This information can be important in improving surgical options with respect to risk and potential benefits in this setting.

ELIGIBILITY:
Inclusion Criteria:

* The patients with clinical diagnosis of PPU underwent laparoscopic repair surgery.

Exclusion Criteria:

* The patients received surgery in an open approach or underwent laparoscopy initially but then intraoperatively converted to laparotomy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: From October 2012 to February 2021, 688 patients presented to the emergency room with a clinical diagnosis of PPU underwent surgery in our hospital. Five hundred and ninety-seven patients were operated in an open approach including 21 patients who were given laparoscopic surgery initially but then intraoperatively converted to laparotomy because the large perforation site cannot be primarily repaired, or the perforation site was difficult to identified or approached. The remaining 91 patients who underwent laparoscopic repair were included in this study.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Short-term outcome with wound infection, pneumonia, leakage, and intraabdominal abscess | Through hospitalization, an average of 8 days
  Complication grading used clavien dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Lien-Cheng Tsao, M.D., Principal Investigator — Changhua Christian Hospital, Changhua, 500, Taiwan